CLINICAL TRIAL: NCT01390831
Title: Renal Denervation in Patients With Uncontrolled Hypertension in Chinese
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second People's Hospital of Chengdu (Other)
Responsible Party: Jian-xiong LIU, The Second People's Hospital of Chengdu
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011SZ0118
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter, Renal Denervation, Ablation (Experimental): Catheter-based renal denervation and maintenance of anti-hypertensive medications
  Interventions: Device: THERMOCOOL® Catheter
- anti-hypertensive medications (No Intervention): Maintenance of anti-hypertensive medications

INTERVENTIONS:
Device: THERMOCOOL® Catheter — Catheter-based renal denervation
  Arms: Catheter, Renal Denervation, Ablation

SUMMARY:
The purpose of this study is to determine whether renal denervation is safe and effective in the treatment of Chinese patients with uncontrolled hypertension.

DETAILED DESCRIPTION:
Prevalence of hypertension is increasing in China.While actually,the controlled rate of hypertension is relatively low,though numerous safe and effective pharmacological therapies are used in clinical practice.Studies confirmed that renal sympathetic nerves contributed to development and perpetuation of hypertension. Previous study has stated that renal denervation was effective and safe in patients with resistant hypertension, while little data is known in Chinese patients. We hypothesis that renal denervation is effective and safe in treatment of Chinese patients with uncontrolled hypertension. This trial plan to recruit 100 patients(Ablation group VS Control group = 1:1) with a follow up duration of 3 years.Patients in ablation group will receive percutaneous renal denervation combined with necessary antihypertension drugs and patients in control group will receive appropriate antihypertension drugs. We aim to explore the long term safety and validity of renal denervation in Chinese patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* a systolic blood pressure of 160mmHg or more and/or a diastolic blood pressure of 90mmHg or more
* receiving and adhering to at least three full doses of appropriate antihypertensive drug regimen
* estimated glomerular filtration rate (eGFR) of ≥45mL/min
* agrees to have the study procedure(s) performed and additional procedures and evaluations
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* secondary hypertension
* renal arterial abnormalities
* has experienced MI, unstable angina pectoris, or CVA within 6 months
* has an implantable cardioverter defibrillator (ICD) or pacemaker, or any other metallic implant which is not compatible with magnetic resonance imaging (MRI)
* requires respiratory support
* patients with sick sinus syndrome
* pregnant woman
* others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Reduction | one year
  To confirm that renal denervation is safe, feasible and effective.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xiong Liu, Principal Investigator — The Second People's Hospital of Chengdu